CLINICAL TRIAL: NCT03375203
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Active- and Placebo-Controlled Polysomnography Study to Evaluate the Efficacy, Safety, and Tolerability of JNJ-42847922 in Subjects With Insomnia Disorder
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of JNJ-42847922 in Participants With Insomnia Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108427; 42847922ISM2005 (Other: Janssen Research & Development, LLC); 2017-000980-33 (EudraCT Number)
Record Dates: First submitted 2017-11-28; First posted 2017-12-15 (Actual); Results first posted 2022-05-23 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Insomnia Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — seltorexant; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Participants will receive matching placebo to JNJ-42847922 as oral capsules at normal study bedtime on Nights 1 through 14.
  Interventions: Drug: Placebo
- JNJ-42847922 5 milligram (mg) (Experimental): Participant will receive JNJ-42847922 5 mg dose as oral capsules at normal study bedtime on Nights 1 through 14.
  Interventions: Drug: JNJ-42847922, 5 mg
- JNJ-42847922 10 mg plus Placebo (Experimental): Participant will receive JNJ-42847922 10 mg as oral capsule and one placebo capsule at normal study bedtime on Nights 1 through 14.
  Interventions: Drug: Placebo; Drug: JNJ-42847922, 10 mg
- JNJ-42847922 20 mg plus Placebo (Experimental): Participant will receive JNJ-42847922 20 mg as oral capsule and one placebo capsule at normal study bedtime on Nights 1 through 14.
  Interventions: Drug: Placebo; Drug: JNJ-42847922, 20 mg
- Zolpidem plus Placebo (Experimental): Participants will receive Zolpidem 5 mg plus one placebo capsule or 10 mg dose as oral capsule at normal study bedtime on Nights 1 through 14.
  Interventions: Drug: Placebo; Drug: Zolpidem

INTERVENTIONS:
Drug: Placebo — Matching placebo will be administered once daily based upon dosing group.
  Arms: JNJ-42847922 10 mg plus Placebo; JNJ-42847922 20 mg plus Placebo; Placebo; Zolpidem plus Placebo
Drug: JNJ-42847922, 5 mg — JNJ-42847922 will be administered as 5 mg (2*2.5 mg capsule) oral capsules once daily.
  Other Names: MIN-202;; Seltorexant
  Arms: JNJ-42847922 5 milligram (mg)
Drug: JNJ-42847922, 10 mg — JNJ-42847922 will be administered as 10 mg oral capsule once daily.
  Other Names: MIN-202;; Seltorexant
  Arms: JNJ-42847922 10 mg plus Placebo
Drug: JNJ-42847922, 20 mg — JNJ-42847922 will be administered as 20 mg oral capsule once daily.
  Other Names: MIN-202;; Seltorexant
  Arms: JNJ-42847922 20 mg plus Placebo
Drug: Zolpidem — Zolpidem will be administered as 5 mg or 10 mg (2*5mg capsule) oral capsule once daily based upon the local labeling information.
  Arms: Zolpidem plus Placebo

SUMMARY:
The purpose of this 2 month phase 2b study is to investigate the dose response of 3 doses of JNJ-42847922 (Seltorexant) (5,10 and 20 mg) compared to placebo and zolpidem on sleep onset and maintenance and to further document safety and tolerability of JNJ-42847922 (Seltorexant) upon multiple (14 days) dose administration in participants with insomnia disorder.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a man or women of non-childbearing potential (WONCBP), 18 to 85 years of age, inclusive, on the day of signing informed consent. A WONCBP is defined as: a).Postmenopausal: A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. b). Permanently sterile: Permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy. c). If reproductive status is questionable, additional evaluation should be considered
* Participant must meet Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5) criteria for insomnia disorder
* Participant must have an Insomnia Severity Index (ISI) total score greater than or equal to (>=) 15 at screening
* Participant must have an self-reported sleep onset latency (sSOL) >=45 minutes and a subjective wake after sleep onset (sWASO) >= 60 minutes on at least 3 nights over any 7-day period during Part 1 of screening, using the Consensus Sleep Diary - Morning Administration (CSD-M), prior to screening polysomnography (PSG) assessments
* Participant must demonstrate a 2-night mean latency to persistent sleep (LPS) of >= 25 minutes (with neither night less than [<] 20 minutes), a 2 night mean wake after sleep onset (WASO) >= 30 minutes, and a 2 night mean total sleep time (TST) less than or equal to (=<) 6.5 hours, with neither night greater than (>) 7 hours
* Participant must be otherwise healthy or present with stable, well-controlled, chronic conditions on the basis of physical examination, medical history, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests performed at screening

Exclusion Criteria:

* Has history of or current clinically significant and/or unstable liver (moderate or severe hepatic impairment [Child-Pugh Score {>=} 7]) or renal insufficiency (severe renal impairment [estimated creatinine clearance below 30 {milliliter per minute} mL/min]; serum creatinine >2 [milligram per deciliter] mg/dL); significant and/or unstable cardiac, vascular, pulmonary (example, acute or severe respiratory failure), gastrointestinal, endocrine, neurologic (example, myasthenia gravis, narcolepsy), hematologic, rheumatologic, immunologic, or metabolic disturbances. Organic brain disease, epilepsy, dementia, narcolepsy, narrow angle glaucoma and known or suspected mental retardation are exclusionary. Any clinically relevant medical condition that is likely to result in deterioration of the participant's condition or affect the participant's safety during the study (eg, medically frail participant with history of hospitalization due to fractures) or could potentially alter the absorption, metabolism, or excretion of the study drug is exclusionary
* Has uncontrolled hypertension (supine systolic blood pressure >150 millimeter of mercury (mm Hg) in adult participants or >160 mm Hg in elderly participants or supine diastolic blood pressure >90 mm Hg, despite diet, exercise, or a stable dose of allowed antihypertensive therapy) at screening or Day 1. (A participant with hypertension may be included if the participant's hypertension has been controlled for at least 3 months prior to screening, and the dosage of any antihypertensive medication has been stable for the past 3 months)
* Has clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening. Participants with non-insulin dependent diabetes mellitus who are adequately controlled (hemoglobin A1c [HbA1c] =< 8 percent [%]) may be eligible to participate if otherwise medically healthy. It is expected that laboratory values will generally be within the normal range, though minor deviations, which are not considered to be of clinical significance to both the investigator and the sponsor's Safety Physician, are acceptable
* Has clinically significant ECG abnormalities at screening or Day 1 prior to randomization defined as:

  1. QT interval corrected according to Fridericia's formula: >= 450 millisecond (msec) (males); >= 470 msec (females).
  2. Evidence of 2nd and 3rd degree atrioventricular block, or 1st degree atrioventricular block with PR interval >210 msec, left bundle branch block.
  3. Features of new ischemia.
  4. Other clinically important arrhythmia
* Has significant hypersomnia not related to night time insomnia (based on clinical judgment of the investigator)
* Regularly naps more than 3 times per week
* Has a current diagnosis or recent history of psychotic disorder, major depressive disorder (MDD), bipolar disorder, or posttraumatic stress disorder, or other psychiatric condition that, in the investigator's opinion, would interfere with the participant's ability to participate in the trial
* Has a current or recent history of serious suicidal ideation within the past 6 months, corresponding to a positive response on item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) for ideation on the Columbia Suicide Severity Rating Scale (C-SSRS), or a history of suicidal behavior within the past year, as validated by the C-SSRS at screening or Day 1. Participants with a prior suicide attempt of any sort, or prior serious suicidal ideation/plan within the past 6 months, should be carefully screened for current suicidal ideation and only participants with non-serious items (1-3 of the suicidal ideation section of the C-SSRS) may be included at the discretion of the investigator
* Has insomnia related to restless leg syndrome (RLS) (defined as periodic leg movement [PLM]-arousal index of >=10 PLM-related electroencephalograph (EEG) arousals per hour of sleep for adult participants or >15 for elderly participants), sleep breathing disorder (defined as an apnea hypopnea index >=10 cumulative apneas and hypopneas per hour of EEG sleep for adult participants or >15 for elderly participants), or parasomnias. These disorders will be ruled out by the first PSG recording during Part 2 of screening
* Has known allergies, hypersensitivity, intolerance, lack of response, or any contraindication to JNJ-42847922 or zolpidem or their excipients
* Plans to father a child while enrolled in this study or within 3 months after the last dose of study drug; and/or, Is pregnant, or breastfeeding, while enrolled in this study or within 1 month after the last dose of study drug

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (56):
- United States (24):
  - Preferred Research Partners, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - California Research Trials DBA Orange Country Research Institute, Anaheim, California
  - Excell Research Inc, Oceanside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Empire Clinical Research, LLC, Upland, California
  - St. Francis Medical Institute, Clearwater, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Sarkis Clinical Trials, Lake City, Florida
  - Innovative Clinical Research Inc, Lauderhill, Florida
  - Suncoast Research Group, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Chicago Research Center, Chicago, Illinois
  - Centennial Medical Group, Elkridge, Maryland
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Gastonia Medical Specialty Clinic, Gastonia, North Carolina
  - Clinical Research of Lake Norman, Mooresville, North Carolina
  - CTI Clinical Trial and Consulting Services, Cincinnati, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Clinical Research of Charleston, Mt. Pleasant, South Carolina
  - FutureSearch Trials of Neurology, LP, Austin, Texas
- Belgium (5):
  - Anima, Alken
  - Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - Universiteit Antwerpen, Wilrijk
- France (4):
  - CHU de Grenoble Hopital Albert Michallon, Isere
  - Hopital de La Croix Rousse, Lyon
  - Hôpital Hôtel Dieu - Paris, Paris
  - Centre Hospitalier Specialisé de Rouffach, Rouffach
- Germany (7):
  - Advanced Sleep Research GmbH, Berlin
  - Emovis GmbH, Berlin
  - Synexus Clinical Research GmbH, Frankfurt
  - CTC North GmbH & Co. KG, Hamburg
  - Synexus Clinical Research GmbH, Sachsen
  - Somni Bene GmbH, Schwerin
  - Klinische Forschung Schwerin GmbH, Schwerin
- Japan (12):
  - SOUSEIKAI PS Clinic, Fukuoka
  - You Ariyoshi Sleep Clinic, Kitakyushu-shi
  - Takedakai Kochi Kagamigawa Hospital, Kochi
  - Kurume University Hospital, Kurume-shi
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Gokeikai Osaka Kaisei Hospital, Osaka
  - Wellness Boyodai Hospital, Otaru-shi
  - Suimin Sogo Care Clinic Yoyogi, Shibuya-ku
  - Shinjuku Research Park Clinic, Shinjuku-ku
  - Sekino Hospital, Toshima-ku
  - Mie University Hospital, Tsu
  - Kaiseikai Kita Shin Yokohama Internal Medicine Clinic, Yokohama
- Poland (4):
  - Centrum Badan Klinicznych PI House sp z o o, Gdansk
  - NZOZ Wielospecjalistyczna Poradnia Lekarska 'Synapsis', Katowice
  - Osrodek Badan Klinicznych CROMED, Poznan
  - EMC Instytut Medyczny SA, Wroclaw

REFERENCES:
- [Derived] Mesens S, Krystal AD, Melkote R, Xu H, Pandina G, Saoud JB, Luthringer R, Savitz A, Drevets WC. Efficacy and Safety of Seltorexant in Insomnia Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2025 Aug 13;82(10):967-76. doi: 10.1001/jamapsychiatry.2025.1999. Online ahead of print. PMID 40802194

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 365 participants were randomized and 364 participants were treated. 1 participant was randomized in error, never received any study drug and was excluded from the analyses. Among 364 treated participants,1 participant randomized to JNJ-42847922 10 mg group, received 5 mg of JNJ-42847922 and was summarized under 5 mg group for safety analyses, and under 10 mg dose group for all other analyses.
Groups:
- Placebo: Participants received matching placebo as 2 oral capsules for 14 consecutive nights from Day 1 to Day 14.
- JNJ-42847922 5 mg: Participants received JNJ-42847922 5 milligrams (mg) dose as two 2.5 mg oral capsules for 14 consecutive nights from Day 1 to Day 14.
- JNJ-42847922 10 mg: Participants received JNJ-42847922 10 mg as one 10 mg oral capsule and one placebo capsule for 14 consecutive nights from Day 1 to Day 14.
- JNJ-42847922 20 mg: Participants received JNJ-42847922 20 mg as one 20 mg oral capsule and one placebo capsule for 14 consecutive nights from Day 1 to Day 14.
- Zolpidem: Participants received Zolpidem 5 mg as one 5 mg capsule plus one placebo capsule or 10 mg Zolpidem as two 5 mg oral capsules for 14 consecutive nights from Day 1 to Day 14.
Period: Overall Study
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Started | 75 | 72 | 74 | 71 | 73
Completed | 69 | 68 | 72 | 69 | 69
Not Completed | 6 | 4 | 2 | 2 | 4
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 3 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 3 | 0 | 1 | 0 | 2
Not completed — Non-compliance with study drug | 1 | 0 | 0 | 0 | 0
Not completed — Randomized, not treated. | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem | Total
Number analyzed (Participants) | 75 | 71 | 74 | 71 | 73 | 364
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (11.49) | 56.9 (13.85) | 57.6 (12.9) | 57.6 (11.88) | 58.5 (12.03) | 57.8 (12.4)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 0 | 0 | 0 | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0 | 0 | 0 | 0
  Adults (18-64 years) | 50 | 45 | 48 | 47 | 48 | 238
  From 65 to 84 years | 25 | 26 | 26 | 24 | 25 | 126
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 48 | 51 | 50 | 52 | 246
  Male | 30 | 23 | 23 | 21 | 21 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 13 | 10 | 7 | 10 | 53
  Not Hispanic or Latino | 62 | 58 | 63 | 64 | 63 | 310
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 1 | 3
  Asian | 8 | 5 | 7 | 4 | 6 | 30
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 3 | 0 | 4
  Black or African American | 11 | 15 | 20 | 18 | 9 | 73
  White | 54 | 49 | 46 | 45 | 57 | 251
  More than one race | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Latency to Persistent Sleep (LPS) as Measured by Polysomnography (PSG) on Night 1
Description: Change in LPS was measured on Night 1 by PSG. LPS is the time in minutes from 'lights out' that marks the starting of total recording time to the first epoch recorded as sleep. The LPS change from baseline on Night 1 was calculated as (LPS at Night 1 minus Baseline LPS). Negative changes in LPS indicated improvement.
Time Frame: Baseline and Night 1
Population: Full analysis set included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 75 | 71 | 73 | 71 | 73
Minutes | -15.24 (78.547) [lower limit 78.547] | -29.92 (49.049) [lower limit 49.049] | -49.49 (53.216) [lower limit 53.216] | -47.69 (48.423) [lower limit 48.423] | -40.74 (54.395) [lower limit 54.395]
Statistical Analysis 1: Comparison: Placebo vs JNJ-42847922 5 mg; Test type: Other; p = 0.346, ANCOVA; Back-transformed Least Square Mean Ratio = 0.88, 90% CI 2-sided [0.70 to 1.10]
Statistical Analysis 2: Comparison: Placebo vs JNJ-42847922 10 mg; Test type: Other; p = 0.001, ANCOVA; Back-transformed Least Square Mean Ratio = 0.64, 90% CI 2-sided [0.51 to 0.81]
Statistical Analysis 3: Comparison: Placebo vs JNJ-42847922 20 mg; Test type: Other; p < 0.001, ANCOVA; Back-transformed Least Square Mean Ratio = 0.51, 90% CI 2-sided [0.41 to 0.64]
Statistical Analysis 4: Comparison: Placebo vs JNJ-42847922 5 mg vs JNJ-42847922 10 mg vs JNJ-42847922 20 mg; Test type: Other; p = 0.000, MCP-mod

2. Secondary Outcome: Change From Baseline in Wake After Sleep Onset (WASO) Over the First 6 Hours as Measured by PSG on Night 1
Description: PSG was used to measure the time to wake after initial sleep onset (WASO) over the first 6 hours on Night 1. Negative changes in WASO indicate improvement.
Time Frame: Baseline and over first 6 hours on Night 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 74 | 71 | 73 | 71 | 73
Minutes | -15.05 (57.485) [lower limit 57.485] | -22.70 (45.904) [lower limit 45.904] | -42.57 (40.011) [lower limit 40.011] | -44.69 (42.823) [lower limit 42.823] | -29.04 (46.779) [lower limit 46.779]

3. Secondary Outcome: Change From Baseline in LPS as Measured by PSG on Night 13
Description: LPS was measured on Night 13 by PSG. LPS is the time in minutes from 'lights out' that marks the starting of total recording time to the first epoch recorded as sleep. Negative changes in LPS indicate improvement.
Time Frame: Baseline and Night 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 69 | 69 | 73 | 69 | 69
Minutes | -23.74 (61.790) [lower limit 61.790] | -27.12 (54.726) [lower limit 54.726] | -53.99 (60.292) [lower limit 60.292] | -41.19 (59.713) [lower limit 59.713] | -30.94 (60.236) [lower limit 60.236]

4. Secondary Outcome: Change From Baseline in WASO Over the First 6 Hours as Measured by PSG on Night 13
Description: PSG was used to measure the time to wake after initial sleep onset (WASO) over the first 6 hours on Night 13. Negative changes in WASO indicate improvement.
Time Frame: Baseline and over first 6 hours on Night 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 68 | 69 | 73 | 68 | 69
Minutes | -17.80 (52.369) [lower limit 52.369] | -14.63 (57.207) [lower limit 57.207] | -30.74 (52.835) [lower limit 52.835] | -38.40 (53.661) [lower limit 53.661] | -20.22 (46.465) [lower limit 46.465]

5. Secondary Outcome: Change From Baseline in Total Sleep Time (TST) as Measured by PSG Over 6 Hours on Nights 1 and 13
Description: TST is defined as the total sleep time in minutes. The total sleep time is the total amount of sleep time scored during the total recording time. Positive changes in TST indicate improvement.
Time Frame: Baseline, Over 6 hours on Nights 1 and 13
Population: Full analysis set included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies number of participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 75 | 71 | 73 | 71 | 73
Minutes
  Night 1 | 25.50 (72.146) | 43.26 (50.771) | 76.47 (50.711) | 80.49 (56.216) | 53.70 (57.688)
  Night 13: number analyzed (Participants) | 69 | 69 | 73 | 69 | 69
  Night 13 | 33.16 (71.488) | 39.80 (66.556) | 66.03 (62.995) | 67.66 (66.254) | 35.84 (64.950)

6. Secondary Outcome: Change From Baseline in Total Sleep Time (TST) as Measured by PSG Over 8 Hours on Nights 1 and 13
Description: as for outcome 5
Time Frame: Baseline, Over 8 hours on Nights 1 and 13
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 75 | 71 | 73 | 71 | 73
Minutes
  Night 1 | 37.03 (86.539) | 47.85 (64.499) | 81.20 (60.607) | 81.07 (71.581) | 63.88 (59.115)
  Night 13: number analyzed (Participants) | 69 | 69 | 73 | 69 | 69
  Night 13 | 38.45 (83.177) | 45.72 (72.640) | 64.84 (77.358) | 64.27 (82.377) | 39.26 (77.773)

7. Secondary Outcome: Change From Baseline in Sleep Efficiency (SE) Measured by PSG on Nights 1 and 13
Description: Sleep efficiency was measured as the total sleep time divided by the total time in bed (that is, the number of hours from the beginning of the Polysomnography recording to the end of the recording) (in percentage). Positive changes in SE indicate improvement.
Time Frame: Baseline, Nights 1 and 13
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of efficient sleep
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 75 | 71 | 73 | 71 | 73
Percentage of efficient sleep
  Night 1 | 7.74 (18.031) | 10.18 (12.818) | 16.92 (12.626) | 16.86 (14.963) | 13.29 (12.317)
  Night 13: number analyzed (Participants) | 69 | 69 | 73 | 69 | 69
  Night 13 | 7.99 (17.322) | 9.51 (15.154) | 13.67 (16.037) | 13.56 (17.199) | 8.27 (16.323)

8. Secondary Outcome: Change From Baseline in Wake After Sleep Onset (WASO) Measured Hourly on Days 1 and 13 From Hour 1 to Hour 8
Description: Polysomnography was used to measure the time to wake after initial sleep onset measured hourly on Day 1 and 13 from Hour 1 to Hour 8. WASO is measured during overnight sleep laboratory (PSG) assessment and defined as the duration of wakefulness from the onset of persistent sleep (that is, 10 consecutive minutes of sleep) over 8 hours of PSG assessment. Negative changes in WASO indicate improvement.
Time Frame: Baseline, Days 1 and 13 (Hours 1 to 8)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 74 | 71 | 73 | 71 | 73
Minutes
  WASO (hour 1): Day 1: number analyzed (Participants) | 43 | 43 | 47 | 50 | 48
  WASO (hour 1): Day 1 | -3.40 (13.074) | -3.55 (10.510) | -3.44 (12.969) | -6.37 (14.213) | -5.40 (12.086)
  WASO (hour 1): Day 13: number analyzed (Participants) | 42 | 41 | 46 | 48 | 45
  WASO (hour 1): Day 13 | 0.43 (12.083) | -4.78 (8.824) | -7.05 (14.569) | -7.47 (13.004) | -4.90 (11.821)
  WASO (hour 2): Day 1: number analyzed (Participants) | 66 | 62 | 66 | 67 | 64
  WASO (hour 2): Day 1 | 1.06 (18.481) | -5.72 (11.817) | -9.62 (16.721) | -10.82 (13.658) | -7.68 (14.812)
  WASO (hour 2):Day 13: number analyzed (Participants) | 61 | 63 | 67 | 63 | 59
  WASO (hour 2):Day 13 | 1.11 (18.504) | -4.12 (14.596) | -9.04 (17.034) | -9.64 (14.963) | -4.37 (16.883)
  WASO (hour 3): Day 1: number analyzed (Participants) | 69 | 69 | 72 | 70 | 71
  WASO (hour 3): Day 1 | -5.57 (18.316) | -3.91 (12.037) | -11.05 (13.272) | -9.64 (13.055) | -9.62 (14.141)
  WASO (hour 3): Day 13: number analyzed (Participants) | 64 | 67 | 71 | 67 | 66
  WASO (hour 3): Day 13 | -5.70 (17.681) | -0.31 (18.562) | -8.10 (12.446) | -6.99 (15.331) | -5.12 (18.140)
  WASO (hour 4): Day 1: number analyzed (Participants) | 72 | 71 | 72 | 71 | 72
  WASO (hour 4): Day 1 | -5.33 (17.109) | -4.73 (13.193) | -9.67 (14.495) | -9.74 (14.727) | -6.23 (16.471)
  WASO (hour 4): Day 13: number analyzed (Participants) | 67 | 69 | 71 | 68 | 67
  WASO (hour 4): Day 13 | -5.49 (18.185) | -3.47 (16.754) | -9.57 (14.483) | -6.21 (14.140) | -7.00 (15.727)
  WASO (hour 5): Day 1: number analyzed (Participants) | 73 | 71 | 73 | 71 | 73
  WASO (hour 5): Day 1 | -3.36 (22.284) | -6.16 (15.820) | -7.53 (14.371) | -7.44 (15.834) | -4.34 (16.150)
  WASO (hour 5): Day 13: number analyzed (Participants) | 68 | 69 | 73 | 69 | 69
  WASO (hour 5): Day 13 | -4.96 (22.597) | -4.06 (20.776) | -5.34 (20.232) | -7.97 (17.016) | -5.03 (16.306)
  WASO (hour 6): Day 1 | -1.06 (17.258) | -4.46 (22.383) | -5.44 (17.510) | -7.78 (18.348) | -1.46 (19.965)
  WASO (hour 6): Day 13: number analyzed (Participants) | 68 | 69 | 73 | 69 | 69
  WASO (hour 6): Day 13 | -4.69 (19.658) | -3.09 (21.426) | 0.56 (22.721) | -7.37 (20.872) | 0.84 (20.768)
  WASO (hour 7): Day 1 | -5.01 (22.247) | -5.71 (19.784) | -3.84 (16.756) | -1.61 (19.349) | -6.15 (13.756)
  WASO (hour 7): Day 13: number analyzed (Participants) | 69 | 69 | 73 | 69 | 69
  WASO (hour 7): Day 13 | -3.57 (21.828) | -4.92 (18.271) | -1.50 (21.145) | 1.16 (23.642) | -0.75 (18.096)
  WASO (hour 8): Day 1 | -7.52 (23.369) | 0.66 (21.311) | -0.65 (22.278) | 1.25 (22.046) | -3.95 (20.149)
  WASO (hour 8): Day 13: number analyzed (Participants) | 69 | 69 | 73 | 69 | 69
  WASO (hour 8): Day 13 | -1.73 (24.898) | -0.63 (20.118) | 1.88 (23.845) | 1.24 (20.858) | -3.22 (22.343)

9. Secondary Outcome: Change From Baseline in Number of Night-time Awakenings (nNAW) Over 6 Hours on Day 1 and 13
Description: PSG was used to measure the number of night-time awakenings over the first 6 hours after initial sleep onset. Negative changes in nNAW indicate improvement.
Time Frame: Baseline, Over 6 hours on Day 1 and 13
Population: FAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies number of participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 74 | 71 | 73 | 71 | 73
awakenings
  Day 1 | -2.08 (6.412) | -0.87 (7.224) | 0.14 (7.385) | -0.94 (9.102) | -1.14 (8.727)
  Day 13: number analyzed (Participants) | 69 | 69 | 73 | 69 | 69
  Day 13 | -2.02 (6.928) | 0.93 (7.769) | -0.40 (8.352) | -2.13 (7.542) | -0.57 (7.803)

10. Secondary Outcome: Change From Baseline in Wake During Total Sleep Period on Day 1 and 13
Description: PSG was used to measure wake time during the total recording period. Negative changes in wake during total sleep period indicate improvement.
Time Frame: Baseline, Day 1 and 13
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 74 | 71 | 73 | 71 | 73
Minutes
  Day 1 | -13.79 (63.082) | -27.47 (58.188) | -49.64 (47.106) | -52.25 (40.828) | -32.36 (53.737)
  Day 13: number analyzed (Participants) | 69 | 69 | 73 | 69 | 69
  Day 13 | -18.83 (59.005) | -19.79 (60.626) | -42.57 (53.867) | -41.95 (64.846) | -20.58 (56.799)

11. Secondary Outcome: Change From Baseline in Wake After Final Awakening on Day 1 and 13
Description: PSG was used to measure the time awake after final awakening to the end of the PSG period. Negative changes in wake after final awakening indicate improvement.
Time Frame: Baseline, Day 1 and 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 74 | 71 | 73 | 71 | 73
Minutes
  Day 1 | -13.63 (50.958) | -0.28 (29.552) | 2.80 (38.492) | 7.21 (45.189) | -5.40 (29.473)
  Day 13: number analyzed (Participants) | 69 | 69 | 73 | 69 | 69
  Day 13 | -5.32 (55.112) | -0.39 (31.519) | 12.42 (62.515) | 5.62 (48.641) | -2.17 (29.376)

12. Secondary Outcome: Change From Baseline in Number of Night-time Awakenings Per Hour (nNAW/hr) on Day 1 and 13
Description: PSG was used to measure number of night time awakenings per hour. Negative changes in nNAW/hr indicate improvement.
Time Frame: Baseline, Day 1 and 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Number of awakenings per hour
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 74 | 71 | 73 | 71 | 73
Number of awakenings per hour
  Day 1 | -0.35 (1.069) | -0.14 (1.204) | 0.02 (1.231) | -0.16 (1.517) | -0.19 (1.455)
  Day 13: number analyzed (Participants) | 69 | 69 | 73 | 69 | 69
  Day 13 | -0.34 (1.155) | 0.16 (1.295) | -0.07 (1.392) | -0.36 (1.257) | -0.10 (1.300)

13. Secondary Outcome: Change From Baseline in Time to First Awakening After Sleep on Day 1 and 13
Description: PSG was used to measure the time to first awakening after sleep onset. Positive changes in time to first awakening after sleep indicate improvement.
Time Frame: Baseline, Day 1 and 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 74 | 71 | 73 | 70 | 73
Minutes
  Day 1 | 12.05 (57.535) | 10.71 (61.015) | 23.11 (73.749) | 53.90 (92.802) | 35.63 (74.617)
  Day 13: number analyzed (Participants) | 69 | 69 | 71 | 68 | 67
  Day 13 | 11.08 (45.714) | 32.13 (70.549) | 33.12 (71.826) | 48.92 (88.909) | 27.55 (75.080)

14. Secondary Outcome: Change From Baseline in Rapid Eye Movement (REM) Duration on Day 1 and 13
Description: PSG was used to measure REM duration (time to first REM period from sleep onset).
Time Frame: Baseline, Day 1 and 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 74 | 71 | 73 | 71 | 73
Minutes
  Day 1 | 10.32 (24.366) | 10.23 (28.891) | 25.12 (29.495) | 23.79 (31.175) | 5.41 (22.381)
  Day 13: number analyzed (Participants) | 69 | 69 | 73 | 69 | 69
  Day 13 | 5.70 (29.875) | 6.40 (25.188) | 17.42 (28.699) | 12.91 (32.051) | 5.97 (28.811)

15. Secondary Outcome: Change From Baseline in Rapid Eye Movement (REM) Latency on Day 1 and 13
Description: PSG was used to measure the REM latency. REM latency was defined as the time to first REM from sleep onset to reaching the first epoch of REM sleep.
Time Frame: Baseline, Day 1 and 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Minute
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 73 | 70 | 73 | 70 | 72
Minute
  Day 1 | -26.60 (82.487) | -38.06 (79.396) | -85.61 (84.380) | -88.36 (76.551) | -42.73 (67.024)
  Day 13: number analyzed (Participants) | 67 | 67 | 72 | 67 | 67
  Day 13 | -26.41 (87.903) | -32.11 (86.623) | -83.89 (83.313) | -73.40 (81.747) | -31.59 (64.953)

16. Secondary Outcome: Percentage of Participants With Sleep-Onset Rapid Eye Movement on Day 1 and 13
Description: PSG was used to measure the sleep-onset REM in participants. REM sleep periods within 15 minutes from sleep onset were measured.
Time Frame: Day 1 and 13
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 75 | 71 | 73 | 71 | 73
percentage of participants
  Day 1 | 1.3 | 4.2 | 9.6 | 14.1 | 0
  Day 13: number analyzed (Participants) | 69 | 69 | 73 | 69 | 69
  Day 13 | 1.4 | 2.9 | 4.1 | 8.7 | 2.9

17. Secondary Outcome: Change From Baseline in Number of Sleep Cycles on Day 1 and 13
Description: PSG was used to measure the number of sleep cycles.
Time Frame: Baseline, Day 1 and 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: sleep cycles
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 75 | 71 | 73 | 71 | 73
sleep cycles
  Day 1 | 0.43 (1.138) | 0.40 (1.006) | 0.97 (1.049) | 0.75 (1.155) | 0.62 (0.941)
  Day 13: number analyzed (Participants) | 69 | 69 | 73 | 69 | 69
  Day 13 | 0.20 (1.222) | 0.41 (1.062) | 0.77 (1.182) | 0.45 (1.219) | 0.32 (0.955)

18. Secondary Outcome: Change From Baseline in Total Time Spent in Non-Rapid Eye Movement Sleep on Day 1 and 13
Description: PSG was used to measure total time spent in non-rapid eye movement sleep stages N1, N2 and N3. Total time spent was sum of N1, N2 and N3. Positive changes in NREM duration indicate improvement.
Time Frame: Baseline, Day 1 and 13
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 75 | 71 | 73 | 71 | 73
Minutes
  Day 1 | 27.87 (68.202) | 37.62 (49.817) | 56.08 (45.218) | 57.29 (54.245) | 58.47 (52.803)
  Day 13: number analyzed (Participants) | 69 | 69 | 73 | 69 | 69
  Day 13 | 32.74 (61.726) | 39.33 (61.524) | 47.41 (59.791) | 51.37 (59.310) | 33.28 (62.466)

19. Secondary Outcome: Change From Baseline in Subjective Sleep Parameters Using Consensus Sleep Diary - Morning Administration (CSD-M) on Days 2 and 14: Self-Reported Sleep-Onset Latency (sSOL), Subjective Wake After Sleep Onset (sWASO), Subjective Total Sleep Time (sTST)
Description: CSD-M is a standardized participant diary based on expert consensus and qualitative participant input to retrieve patient reported subjective sleep parameters related to prior night's sleep. CSD-M parameters analyzed includes: sSOL, sTST, sWASO. Negative change in sSOL, sWASO indicate improvement. Positive change in sTST indicates improvement.
Time Frame: Baseline, Days 2 and 14
Population: FAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 71 | 66 | 68 | 69 | 68
Minutes
  sSOL: Day 2 | 15.20 (61.761) | -3.99 (46.858) | -16.49 (42.699) | -27.60 (34.456) | -24.98 (30.395)
  sSOL: Day 14: number analyzed (Participants) | 63 | 64 | 67 | 65 | 66
  sSOL: Day 14 | 10.92 (68.201) | -8.81 (45.936) | -31.33 (36.888) | -33.93 (37.274) | -14.53 (53.705)
  sWASO: Day 2: number analyzed (Participants) | 69 | 64 | 68 | 64 | 61
  sWASO: Day 2 | 0.81 (75.475) | -5.47 (61.067) | -18.54 (51.301) | -13.28 (48.225) | -15.99 (84.549)
  sWASO : Day 14: number analyzed (Participants) | 59 | 61 | 64 | 62 | 60
  sWASO : Day 14 | -5.60 (55.955) | -18.25 (56.719) | -25.20 (58.872) | -20.16 (65.568) | -17.56 (51.007)
  sTST: Day 2 | -12.64 (96.051) | 4.90 (92.105) | 29.25 (67.934) | 34.50 (76.904) | 37.07 (71.297)
  sTST: Day 14: number analyzed (Participants) | 63 | 64 | 67 | 65 | 66
  sTST: Day 14 | 3.30 (89.019) | 29.34 (83.772) | 36.79 (88.379) | 45.35 (81.983) | 27.68 (90.387)

20. Secondary Outcome: Change From Baseline in Subjective Sleep Parameters Using Consensus Sleep Diary - Morning Administration (CSD-M) on Days 2 and 14: Subjective Refreshed Feeling on Waking (sFRESH) and Subjective Quality of Sleep (sQUAL)
Description: The CSD-M is a standardized participant diary based on expert consensus and qualitative participant input to retrieve patient reported subjective sleep parameters related to the prior night's sleep. Sleep quality and how well rested participants felt at awaking are rated on a 5-point Likert scale ranging from 1 (very poor) to 5 (very good). Higher ratings indicate better sleep quality (sQUAL) and more refreshing/restorative quality of sleep (sFRESH). CSD-M parameters analyzed includes: sFRESH and sQUAL. Positive change in sFRESH and sQUAL indicates improvement.
Time Frame: Baseline, Days 2 and 14
Population: Full analysis set included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 71 | 66 | 68 | 69 | 68
Units on a Scale
  sFRESH: Day 2 | 0.07 (0.930) | 0.14 (0.865) | 0.34 (0.852) | 0.58 (1.050) | 0.41 (0.876)
  sFRESH: Day 14: number analyzed (Participants) | 63 | 64 | 67 | 65 | 66
  sFRESH: Day 14 | 0.26 (0.826) | 0.39 (1.081) | 0.51 (1.005) | 0.59 (1.018) | 0.41 (1.051)
  sQUAL: Day 2 | 0.11 (0.995) | 0.14 (1.054) | 0.49 (0.896) | 0.49 (1.091) | 0.66 (0.818)
  sQUAL: Day 14: number analyzed (Participants) | 63 | 64 | 67 | 65 | 66
  sQUAL: Day 14 | 0.26 (1.024) | 0.43 (1.172) | 0.79 (1.189) | 0.67 (1.159) | 0.52 (1.084)

21. Secondary Outcome: Change From Baseline in Subjective Sleep Parameters Using Consensus Sleep Diary - Morning Administration (CSD-M) on Days 2 and 14: Number of Nighttime Awakenings (s-nNAW)
Description: CSD-M is a standardized participant diary based on expert consensus and qualitative participant input to retrieve patient reported subjective sleep parameters related to the prior night's sleep. CSD-M parameters analyzed include: s-nNAW. Negative change in s-nNAW indicate improvement.
Time Frame: Baseline, Days 2 and 14
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 71 | 66 | 68 | 69 | 68
awakenings
  Day 2 | 0.64 (2.197) | 0.21 (1.465) | 0.49 (1.465) | 0.27 (1.418) | 0.38 (6.076)
  Day 14: number analyzed (Participants) | 63 | 64 | 67 | 65 | 66
  Day 14 | 0.10 (1.234) | 0.04 (1.580) | 0.05 (1.320) | -0.02 (1.175) | -0.22 (1.376)

22. Secondary Outcome: Change From Baseline in Sleep Disturbance as Measured by Patient Reported Outcome Measurement Information System - Sleep Disturbance (PROMIS-SD) Total Score on Days 8 and 14
Description: PROMIS Sleep Disturbance (PROMIS-SD) Short Form subscale consists of a static 8-item questionnaire. Using a recall period of the past 7 days, it assesses the concepts of sleep initiation (2 items), quality of sleep (3 items), early morning feelings (2 items) and worrying about sleep (1 item). Each question has 5 response options ranging in value from 1 to 5. To find the total raw score for a short form with all questions answered, sum the values of the response to each question and a total score ranges from 8 to 40. Lower scores indicate less sleep disturbance. Negative changes in scores indicate improvement.
Time Frame: Baseline, Days 8 and 14
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Unit on a Scale
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 63 | 60 | 66 | 63 | 66
Unit on a Scale
  Day 8: number analyzed (Participants) | 59 | 55 | 59 | 58 | 58
  Day 8 | -4.9 (6.81) | -9.0 (7.13) | -9.2 (7.17) | -9.6 (8.16) | -8.3 (7.31)
  Day 14 | -5.7 (7.75) | -10.8 (7.64) | -10.3 (7.39) | -9.5 (7.93) | -10.1 (8.06)

23. Secondary Outcome: Change From Baseline in Impairment as Measured by Patient Reported Outcome Measurement Information System - Sleep Related Impairment (PROMIS-SRI) Total Score on Days 8 and 14
Description: PROMIS-Sleep Related Impairment (PROMIS-SRI) scale consists of 8 items to evaluate daytime consequences of functioning 5-point Likert scale ranging from 1 to 5. PROMIS-SRI measures self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours, and perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. Each question has five response options ranging in value from 1 to 5. To find total raw score (which range from 8 to 40) with all questions answered, sum values of response to each question. Higher score indicates greater sleep impairment.
Time Frame: Baseline, Days 8 and 14
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 61 | 59 | 63 | 62 | 65
Units on a Scale
  Day 8: number analyzed (Participants) | 57 | 54 | 55 | 51 | 54
  Day 8 | -4.0 (6.56) | -7.0 (6.15) | -5.5 (6.55) | -8.8 (7.09) | -4.9 (6.98)
  Day 14 | -5.2 (6.88) | -9.1 (6.53) | -6.3 (6.94) | -7.8 (6.98) | -7.4 (6.35)

24. Secondary Outcome: Change From Baseline in Participant's Assessment of Insomnia Severity Using the Patient Global Impression - Severity (PGI-S) Scale Score on Day 14
Description: The PGI-S is a self-reported scale to measure severity of illness using a 6-point scale ranging from 1 to 6, (1=no insomnia, 2=very mild, 3=mild, 4=moderate, 5=severe, 6=very severe). Considering all aspects of insomnia, participants rated their severity on the PGI-S scale. Negative changes in scores indicate improvement.
Time Frame: Baseline and Day 14
Population: FAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Unit on a Scale
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 59 | 59 | 65 | 62 | 65
Unit on a Scale | 0.00 (-5.0) [-5.0 to 2.0] | -1.00 (-4.0) [-4.0 to 2.0] | -1.00 (-4.0) [-4.0 to 1.0] | -1.00 (-5.0) [-5.0 to 1.0] | -1.00 (-4.0) [-4.0 to 1.0]

25. Secondary Outcome: Participant's Assessment of Improvement in Insomnia Using the Patient Global Impression - Improvement (PGI-I) Scale Score on Day 14
Description: PGI-I is a self-reported scale to measure improvement in illness using a 7-point scale ranging from 1 to 7, (1=very much improved, 2=much improved, 3=improved [just enough to make a difference], 4=no change, 5=worse [just enough to make a difference], 6=much worse, 7=very much worse). Negative changes in scores indicate improvement.
Time Frame: Baseline and Day 14
Population: as for outcome 24
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 60 | 62 | 69 | 65 | 67
Units on a Scale | 3.00 (0.0) [0.0 to 5.0] | 2.00 (0.0) [0.0 to 5.0] | 2.00 (0.0) [0.0 to 4.0] | 2.00 (0.0) [0.0 to 4.0] | 2.00 (0.0) [0.0 to 5.0]

26. Secondary Outcome: Percentage of Participants Who Achieved Response Based on Insomnia Severity Index (ISI) Total Score on Day 14 - Observed Case
Description: Percentage of participants who achieved at least 50% reduction from baseline in ISI total score (responders) were reported. It is a 7-item questionnaire assessing nature, severity, impact of insomnia. Dimensions evaluated: severity of sleep onset, sleep maintenance, early morning awakening problems; sleep dissatisfaction; interference of sleep problem with daytime functioning; noticeability of sleep problems; distress caused by sleep difficulties. 5-point Likert scale (0-4) was used to rate each item, Scores are summed for a total score which ranges from 0-28. Negative changes in scores indicate improvement. ISI total score is the sum of all item scores. Total score interpreted insomnia as follows: absence (0-7); sub-threshold (8-14); moderate (15-21); severe (22-28).
Time Frame: Day 14
Population: FAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies number participants evaluable for this outcome measure. Participants with missing values at a given time point were excluded from frequency calculation for that time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 69 | 69 | 73 | 69 | 70
percentage of participants | 23.2 | 42.0 | 31.5 | 34.8 | 42.9

27. Secondary Outcome: Percentage of Participants Who Achieved Remission Based on Insomnia Severity Index (ISI) Total Score on Day 14 - Observed Case
Description: Percentage of participants with remission of insomnia symptom defined as, total score of <= 10 on ISI scale. ISI is 7-item questionnaire assessing nature, severity, impact of insomnia. Dimensions evaluated are: severity of sleep onset, sleep maintenance, early morning awakening problems; sleep dissatisfaction; interference of sleep problem with daytime functioning; noticeability of sleep problems by others; distress caused by sleep difficulties. 5-point Likert scale (0-4) is used to rate each item. ISI total score is the sum of all item scores. ISI total score is the sum of all item scores. Scores are summed for a total score which ranges from 0-28 and interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); severe insomnia (22-28).
Time Frame: Day 14
Population: FAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Participants with missing values at a given time point are excluded from the frequency calculation for that time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 69 | 69 | 73 | 69 | 70
percentage of participants | 24.6 | 43.5 | 37.0 | 39.1 | 50.0

28. Secondary Outcome: Change From Baseline in Clinician's Assessment of Insomnia Severity Using the Clinical Global Impression - Severity (CGI-S) Score on Day 14
Description: The CGI-S is a 7-point scale to measure severity of illness (1=normal [not at all ill], 2=borderline ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, 7=among the most extremely ill participants). Higher score indicates more severity. Negative changes in scores indicate improvement.
Time Frame: Baseline and Day 14
Population: as for outcome 24
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 69 | 69 | 73 | 69 | 70
Units on a scale | 0.0 [-5 to 1] | -1.0 [-5 to 3] | -1.0 [-5 to 2] | -1.0 [-5 to 1] | -1.0 [-5 to 0]

29. Secondary Outcome: Change From Baseline in Clinician's Assessment of Insomnia Improvement Using Clinical Global Impression-Improvement (CGI-I) Score on Day 14
Description: The CGI-I is a 7-point scale to measure improvement in illness using a 7-point scale ranging from 1 to 7 (1=very much improved, 2=much improved, 3=minimally improved, 4=no change from baseline, 5=minimally worse, 6=much worse, 7=very much worse). Higher score indicates more severity. Negative changes in scores indicate improvement.
Time Frame: Baseline and Day 14
Population: as for outcome 24
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 69 | 69 | 73 | 69 | 70
Units on a Scale | 3.0 [1 to 5] | 3.0 [1 to 5] | 3.0 [1 to 4] | 3.0 [1 to 5] | 2.0 [1 to 5]

30. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) as a Measure of Safety and Tolerability
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Treatment-emergent adverse events are adverse events with an onset date occurring at or after the initial administration of study drug through the Day 17 telephone contact date, or the day of last dose plus 3 days for participants without the Day 17 telephone contact date.
Time Frame: Up to Day 17
Population: Safety analysis set (SAS) included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. One participant who was randomized to JNJ-42847922 10 mg dose group received 5 mg of JNJ-42847922. This participant was summarized under the 5 mg dose group for safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 75 | 72 | 73 | 71 | 73
Participants | 37 | 29 | 23 | 21 | 31

31. Secondary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events and Events of Special Interest
Description: Treatment-emergent serious adverse events are serious adverse events with an onset date occurring at or after the initial administration of study drug through the Day 17 telephone contact date, or the day of last dose plus 3 days for participants without the Day 17 telephone contact date. Events of special interest included: Cataplexy; Sleep paralysis; Complex sleep-related behaviors such as confusional arousals, somnambulism (sleep walking), sleep terrors, bruxism (teeth grinding), sleep sex, sleep related eating disorder, sleep behavior disorder, and catathrenia (REM-associated end-inspiratory apnea/breath holding); Abnormal dreams; Falls.
Time Frame: Up to Day 17
Population: SAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. One participant who was randomized to JNJ-42847922 10 mg dose group received 5 mg of JNJ-42847922. This participant was summarized under the 5 mg dose group for safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 75 | 72 | 73 | 71 | 73
Participants
  Treatment-emergent Serious AE | 0 | 0 | 0 | 1 | 1
  Events of Special Interest | 2 | 1 | 2 | 1 | 4

32. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs and Physical Abnormalities
Description: Clinically significant vital signs (pulse, supine and standing blood pressure (systolic and diastolic), and oral, temperature) and physical abnormalities (body weight) were reported. Abnormally low parameters included pulse (bpm)- decrease value from baseline greater than or equal to (>=) 15 to <=50; Systolic BP (mmHg [Millimeter of mercury])- decrease value from baseline >=20 to <=90; Diastolic BP- decrease value from baseline >=15 to <=50; weight (Kilogram[Kg])- decrease from baseline >=7%; Body temperature (Celsius [C])- <35.5. Abnormally high parameters included pulse- increase value from baseline >=15 to >=100; Systolic BP(mmHg)- increase from baseline of >=20 to >=180; Diastolic BP- increase value from baseline >=15 to >=105; weight(Kg)- increase from baseline of >=7%; body temperature (C)- >37.5.
Time Frame: Up to Day 15
Population: SAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. One participant who was randomized to JNJ-42847922 10 mg dose group received 5 mg of JNJ-42847922. This participant was summarized under the 5 mg dose group for safety analyses. Here, 'n' (number analyzed) signifies number of participants who were evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 75 | 72 | 73 | 71 | 73
Participants
  Supine Pulse Rate: Abnormally low | 2 | 2 | 2 | 3 | 0
  Supine Pulse Rate: Abnormally high | 1 | 0 | 0 | 0 | 1
  Standing Pulse Rate: Abnormally low | 1 | 0 | 0 | 1 | 1
  Standing Pulse Rate: Abnormally high | 8 | 7 | 3 | 6 | 11
  Supine Systolic BP: Abnormally low | 3 | 0 | 3 | 2 | 2
  Supine Systolic BP: Abnormally high | 1 | 0 | 0 | 0 | 0
  Standing Systolic BP: Abnormally low | 2 | 1 | 1 | 3 | 5
  Standing Systolic BP: Abnormally high | 2 | 0 | 0 | 0 | 0
  Supine Diastolic BP: Abnormally low | 2 | 0 | 0 | 0 | 4
  Supine Diastolic BP: Abnormally high | 0 | 1 | 0 | 0 | 1
  Standing Diastolic BP: Abnormally low | 0 | 1 | 0 | 1 | 0
  Standing Diastolic BP: Abnormally high | 0 | 0 | 0 | 0 | 1
  Temperature: Abnormally low | 2 | 3 | 0 | 3 | 2
  Temperature: Abnormally high | 1 | 0 | 0 | 2 | 1
  Weight: Abnormally low: number analyzed (Participants) | 69 | 70 | 71 | 69 | 71
  Weight: Abnormally low | 0 | 0 | 0 | 0 | 0
  Weight: Abnormally high: number analyzed (Participants) | 69 | 70 | 71 | 69 | 71
  Weight: Abnormally high | 2 | 0 | 0 | 1 | 0

33. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Twelve-lead ECGs were recorded in a supine position and different ECG intervals (Respiratory rate [RR], PR, time for ventricular depolarization [QRS], and total time from ventricular depolarization to complete repolarization [QT]) and heart rate was measured. This included heart rate:<=50 beats per minute (bpm) and >=100 bpm; PR interval <=120 millisecond (msec) and >=200 msec; QRS interval: <=60 msec and >=120 msec; QT interval:<=200 msec and >=500 msec.
Time Frame: Up to Day 14
Population: SAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies number of participants who were evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 74 | 70 | 71 | 68 | 71
Participants
  Heart rate: <=50 bpm | 10 | 7 | 5 | 6 | 6
  Heart rate:>=100 bpm | 0 | 0 | 0 | 0 | 0
  PR interval: <=120 msec: number analyzed (Participants) | 74 | 69 | 71 | 68 | 71
  PR interval: <=120 msec | 0 | 0 | 0 | 1 | 0
  PR interval: >=200 msec: number analyzed (Participants) | 74 | 69 | 71 | 68 | 71
  PR interval: >=200 msec | 4 | 4 | 4 | 2 | 7
  QRS interval: <=60 msec | 0 | 0 | 0 | 0 | 0
  QRS interval: >=120 msec | 0 | 0 | 0 | 0 | 0
  QT interval: <=200 msec | 0 | 0 | 0 | 0 | 0
  QT interval: >=500 msec | 1 | 0 | 0 | 1 | 0

34. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Number of participants with clinically significant laboratory abnormalities were reported. Blood samples for serum chemistry (albumin, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, bicarbonate, calcium, chloride, creatine Kinase, gamma glutamyl transferase, lactate dehydrogenase, phosphate, potassium, sodium), and urinalysis (bilirubin, protein) were collected for clinical laboratory testing.
Time Frame: Up to Day 15
Population: Analysis population was SAS. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here,'n' (number analyzed) signifies number of participants who were evaluable for specified categories. 1 participant who was randomized to JNJ-42847922 10 mg dose group received 5 mg of JNJ-42847922.This participant was summarized under the 5 mg dose group for safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 69 | 70 | 71 | 68 | 71
Participants
  Alanine Aminotransferase: Abnormally high: number analyzed (Participants) | 69 | 70 | 69 | 67 | 71
  Alanine Aminotransferase: Abnormally high | 0 | 0 | 0 | 0 | 0
  Albumin: Abnormally low | 0 | 0 | 0 | 0 | 0
  Albumin: Abnormally high | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase: Abnormally high: number analyzed (Participants) | 69 | 70 | 70 | 68 | 71
  Alkaline Phosphatase: Abnormally high | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase: Abnormally high: number analyzed (Participants) | 69 | 70 | 69 | 67 | 71
  Aspartate Aminotransferase: Abnormally high | 0 | 0 | 0 | 0 | 0
  Bicarbonate: Abnormally low: number analyzed (Participants) | 69 | 70 | 69 | 67 | 71
  Bicarbonate: Abnormally low | 0 | 0 | 0 | 0 | 0
  Bicarbonate: Abnormally high: number analyzed (Participants) | 69 | 70 | 69 | 67 | 71
  Bicarbonate: Abnormally high | 0 | 0 | 0 | 0 | 0
  Bilirubin: Abnormally high: number analyzed (Participants) | 69 | 70 | 69 | 67 | 71
  Bilirubin: Abnormally high | 0 | 0 | 0 | 0 | 0
  Calcium: Abnormally low: number analyzed (Participants) | 69 | 70 | 70 | 68 | 71
  Calcium: Abnormally low | 0 | 0 | 0 | 0 | 0
  Calcium: Abnormally high: number analyzed (Participants) | 69 | 70 | 70 | 68 | 71
  Calcium: Abnormally high | 0 | 0 | 0 | 0 | 0
  Chloride: Abnormally low: number analyzed (Participants) | 69 | 70 | 70 | 68 | 71
  Chloride: Abnormally low | 1 | 0 | 0 | 0 | 0
  Chloride: Abnormally high: number analyzed (Participants) | 69 | 70 | 70 | 68 | 71
  Chloride: Abnormally high | 0 | 0 | 0 | 0 | 0
  Creatine Kinase: Abnormally high: number analyzed (Participants) | 69 | 70 | 69 | 67 | 71
  Creatine Kinase: Abnormally high | 0 | 1 | 0 | 0 | 0
  Creatinine: Abnormally high: number analyzed (Participants) | 69 | 70 | 70 | 68 | 71
  Creatinine: Abnormally high | 0 | 1 | 0 | 0 | 0
  Direct Bilirubin: Abnormally high: number analyzed (Participants) | 68 | 70 | 69 | 66 | 70
  Direct Bilirubin: Abnormally high | 0 | 0 | 0 | 0 | 0
  Gamma Glutamyl Transferase: Abnormally high: number analyzed (Participants) | 69 | 70 | 70 | 68 | 71
  Gamma Glutamyl Transferase: Abnormally high | 0 | 0 | 0 | 0 | 0
  Lactate Dehydrogenase: Abnormally high: number analyzed (Participants) | 62 | 68 | 65 | 65 | 64
  Lactate Dehydrogenase: Abnormally high | 0 | 0 | 1 | 0 | 0
  Phosphate: Abnormally low | 0 | 0 | 0 | 0 | 0
  Phosphate: Abnormally high | 0 | 0 | 0 | 0 | 0
  Potassium: Abnormally low: number analyzed (Participants) | 69 | 70 | 70 | 68 | 71
  Potassium: Abnormally low | 0 | 0 | 0 | 0 | 0
  Potassium: Abnormally high: number analyzed (Participants) | 69 | 70 | 70 | 68 | 71
  Potassium: Abnormally high | 0 | 0 | 3 | 1 | 2
  Protein: Abnormally low: number analyzed (Participants) | 69 | 70 | 70 | 68 | 71
  Protein: Abnormally low | 0 | 1 | 0 | 0 | 0
  Sodium: Abnormally low: number analyzed (Participants) | 69 | 70 | 70 | 68 | 71
  Sodium: Abnormally low | 0 | 0 | 0 | 0 | 0
  Sodium: Abnormally high: number analyzed (Participants) | 69 | 70 | 70 | 68 | 71
  Sodium: Abnormally high | 0 | 0 | 0 | 0 | 0

35. Secondary Outcome: Number of Participants With Suicidal Ideation and Behavior as Determined by Columbia Suicide Severity Rating Scale (C-SSRS) Score
Description: C-SSRS is a questionnaire designed to solicit occurrence, severity, frequency of suicidal ideation/behaviors using following scores: Suicidal Ideation-1:Wish to be Dead; 2:Non-specific Active Suicidal Thoughts; 3:Active Suicidal Ideation with Any Methods without Intent to Act; 4:Active Suicidal Ideation with Some Intent to Act; 5:Active Suicidal Ideation with Specific Plan/Intent; Suicidal Behavior-6:Preparatory Acts; 7:Aborted Attempt; 8:Interrupted Attempt; 9:Actual Attempt; 10:Completed Suicide. If no events qualify for score of 1-10, score 0 indicate "no event that can be assessed on basis of C-SSRS". Higher scores= greater severity.
Time Frame: Day 14
Population: SAS included all participants who were randomly assigned to drug and received at least 1 dose of drug. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure. 1 participant who was randomized to JNJ-42847922 10 mg dose group received 5 mg of JNJ-42847922 and was summarized under 5 mg dose group for safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 69 | 70 | 72 | 69 | 70
Participants
  Score 0: No Event | 69 | 70 | 72 | 69 | 70
  Score 1: Wish to be Dead | 0 | 0 | 0 | 0 | 0
  Score 2: Non-Specific Active Suicidal Thoughts | 0 | 0 | 0 | 0 | 0
  Score 3: Suicidal Ideation Without Plan and Intent | 0 | 0 | 0 | 0 | 0
  Score 4: Suicidal Ideation Intent to Act Without Plan | 0 | 0 | 0 | 0 | 0
  Score 5: Suicidal Ideation With Plan and Intent | 0 | 0 | 0 | 0 | 0
  Score 6: Preparatory Acts or Behavior | 0 | 0 | 0 | 0 | 0
  Score 7: Aborted Attempt | 0 | 0 | 0 | 0 | 0
  Score 8: Interrupted Attempt | 0 | 0 | 0 | 0 | 0
  Score 9: Actual Attempt | 0 | 0 | 0 | 0 | 0
  Score 10: Completed Suicide | 0 | 0 | 0 | 0 | 0

36. Secondary Outcome: Change From Baseline in Karolinska Sleepiness Scale (KSS) Total Score on Days 2 and 14
Description: The KSS is a patient reported assessment of level of drowsiness at the time of scale administration. This scale is focused mainly on the propensity to fall asleep and has a high validity in measuring sleepiness. It consists of a single item assessed on 9-point Likert scale with response options from: 1=very alert to 9=very sleepy (fighting sleep). Negative changes indicate improvement.
Time Frame: Baseline, Days 2 and 14
Population: Analysis population was SAS. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies number of participants who were evaluable at specified time points. One participant who was randomized to JNJ-42847922 10 mg dose group received 5 mg of JNJ-42847922. This participant was summarized under the 5 mg dose group for safety analyses.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 66 | 62 | 65 | 59 | 67
Units on a Scale
  Day 2: number analyzed (Participants) | 66 | 61 | 65 | 59 | 67
  Day 2 | 0.3 (1.75) | -0.4 (1.86) | -0.2 (1.42) | -0.5 (1.86) | -0.4 (1.68)
  Day 14: number analyzed (Participants) | 63 | 62 | 62 | 59 | 65
  Day 14 | 0.1 (1.82) | -0.8 (2.15) | -0.6 (1.72) | -0.7 (1.90) | -0.7 (2.01)

37. Secondary Outcome: Postural Stability Measured by Ataxiameter
Description: The body sway meter allows measurement of body movements in a single plane, providing a measure of postural stability. Body sway was measured using an ataxiameter. Participants were instructed to wear a pair of thin socks for each session. Before starting a measurement, participants were asked to stand still and comfortable, with their feet approximately 10 centimeters (cm) apart and their hands in a relaxed position alongside the body and eyes closed. The total period of body sway measurement was 2 minutes.
Time Frame: Day 14 (morning)
Population: SAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure. One participant who was randomized to JNJ-42847922 10mg dose group received 5 mg of JNJ-42847922. This participant was summarized under the 5 mg dose group for safety analyses.
Measure: Mean (Standard Deviation); unit: 1/3 Degree Angle of Arc
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 66 | 66 | 69 | 67 | 69
1/3 Degree Angle of Arc | -0.06 (17.15) | 3.14 (16.14) | -0.87 (15.62) | -0.25 (14.71) | 1.65 (14.11)

38. Secondary Outcome: Change From Baseline in Power of Attention as Measured by a Computerized Battery of Cognitive Tests on Day 14 (Morning)
Description: Power of Attention is a combination of the speed scores from the three tests of attention, and is established to reflect the ability to focus attention and to process information. Power of Attention was calculated from the sum of the reaction time measured from the attentional tasks (Simple Reaction Time, Choice Reaction Time and Digit Vigilance Speed). Score ranges from 450 milliseconds - 61500 milliseconds. A low score reflects a fast reaction time and a high intensity of concentration.
Time Frame: Baseline and Day 14 (Morning)
Population: SAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure. One participant who was randomized to JNJ-42847922 10 mg dose group received 5 mg of JNJ-42847922. This participant was summarized under the 5 mg dose group for safety analyses.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 67 | 66 | 68 | 67 | 69
milliseconds (ms) | 35.88 (125.43) | 48.59 (137.75) | 67.09 (257.67) | 37.07 (124.23) | 35.38 (189.99)

39. Secondary Outcome: Change From Baseline in Continuity of Attention as Measured by a Computerized Battery of Cognitive Tests on Day 14 (Morning)
Description: Continuity of attention is a measure of sustained attention, combining (summed) accuracy and error measures from the choice reaction time and digit vigilance tasks. The number of correct responses (out of 50) for choice reaction time was added to the total number of targets correctly identified (out of 45) digit vigilance minus the number of false alarms (total score of -45 to 95). A high score reflects someone able to keep his/her mind on a single task for a prolonged period. A negative change from baseline reflects impairment compared to baseline.
Time Frame: Baseline and Day 14 (Morning)
Population: SAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies number of participants evaluable for this endpoint. One participant who was randomized to JNJ-42847922 10 mg dose group received 5 mg of JNJ-42847922. This participant was summarized under the 5 mg dose group for safety analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 67 | 66 | 68 | 67 | 69
units on a scale | 0.36 (5.31) | -0.20 (3.16) | -1.37 (6.35) | 0.10 (5.05) | -0.39 (5.14)

40. Secondary Outcome: Change From Baseline in Quality of Working Memory as Measured by a Computerized Battery of Cognitive Tests on Day 14 (Morning)
Description: Quality of working memory is a combination of the scores from Spatial Working Memory and Numeric Working Memory tasks, and is established to reflect the ability to temporarily hold numeric and spatial information in memory. Sum of Spatial and Numeric Working Memory sensitivity indices (SI) (accuracy) was used to calculate the quality of working memory. The quality of working memory score was calculated from formulae that combined the accuracy scores for the original as well as the new (distractor) stimuli. The range for both the numeric working memory and spatial working memory tasks SI are -1 to 1. Smaller scores reflect poorer ability (poorer quality of working memory),larger scores reflect better ability (better quality of working memory). Total score is the sum of Spatial Working Memory and Numeric Working Memory (ranges from -2 to 2). Smaller scores reflect poorer ability (poorer quality of working memory), larger scores reflect better ability (better quality of working memory.
Time Frame: Baseline and Day 14 (Morning)
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 67 | 65 | 68 | 67 | 69
Units on scale | 0.00 (0.35) | -0.03 (0.28) | -0.02 (0.41) | -0.04 (0.29) | 0.05 (0.28)

41. Secondary Outcome: Change From Baseline in Quality of Episodic Secondary Memory as Measured by a Computerized Battery of Cognitive Tests on Day 14 (Morning)
Description: Quality of episodic secondary memory is calculated from the sum of 4 tests: Immediate and delayed word recall, and word and picture recognition, and ranges from -200 to 400. A high score reflects a good ability to store, hold and retrieve information of an episodic nature (that is an event or a name) and a negative change from baseline reflects impairment compared to baseline.
Time Frame: Baseline and Day 14 (Morning)
Population: SAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. One participant who was randomized to JNJ-42847922 10 mg dose group received 5 mg of JNJ-42847922. This participant is summarized under the 5 mg dose group. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 66 | 65 | 68 | 66 | 67
units on scale | -22.84 (53.73) | -23.15 (46.02) | -33.58 (48.82) | -25.45 (56.37) | -37.96 (55.94)

42. Secondary Outcome: Change From Baseline in Speed of Memory as Measured by a Computerized Battery of Cognitive Tests on Day 14 (Morning)
Description: The sum of the speed measures from the two working memory tasks (Spatial and Numeric) and the two recognition tasks (Word and Picture). Speed of Memory combines reaction times from Spatial Working Memory (range:150 to 30000 millisecond [ms]), Numeric Working Memory (150 to 30000 ms), Word Recognition (250 to 30000 ms) and Picture recognition (250 to 30000 ms) tasks. The total reaction time (sum of above 4 reaction times) measures memory retrieval speed which ranges from 800 to 120000 ms. Slower reaction time reflect poorer ability and faster reaction time reflect better ability.
Time Frame: Baseline and Day 14 (Morning)
Population: SAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. One participant who was randomized to JNJ-42847922 10 mg dose group received 5 mg of JNJ-42847922. This participant was summarized under the 5 mg dose group for safety analyses. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 67 | 65 | 68 | 67 | 69
millisecond | -104.75 (787.74) | 258.38 (719.56) | 7.57 (806.27) | -65.67 (761.77) | -83.70 (1060.38)

43. Secondary Outcome: Change in Subjective Sleep Parameters From Day 14 as Compared to Day 17 as Measured by the Consensus Sleep Diary-Morning Administration (CSD-M):Self-Reported Sleep-Onset Latency (sSOL), Subjective Wake After Sleep Onset (sWASO) and sTST
Description: CSD-M is a standardized participant diary based on expert consensus and qualitative participant input to retrieve patient reported subjective sleep parameters related to prior night's sleep. Negative change in sSOL, sWASO indicate improvement and positive change in Subjective Total Sleep Time (sTST) indicates improvement.
Time Frame: Day 14 to Day 17
Population: FAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies number of participants who were evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 63 | 58 | 57 | 56 | 58
Minutes
  sSOL | -20.56 (74.145) | -4.83 (43.769) | 9.67 (29.798) | 15.55 (32.327) | 9.57 (72.253)
  sWASO: number analyzed (Participants) | 57 | 51 | 52 | 51 | 51
  sWASO | -12.39 (57.711) | -0.76 (66.663) | -2.13 (41.505) | -10.80 (63.672) | 3.76 (58.805)
  sTST | 30.95 (101.367) | 13.07 (102.093) | 6.96 (96.664) | 19.71 (66.447) | -7.95 (102.183)

44. Secondary Outcome: Change in Subjective Sleep Parameters From Day 14 as Compared to Day 17 Using Consensus Sleep Diary-Morning Administration: Subjective Refreshed Feeling on Waking (sFRESH) and Subjective Quality of Sleep (sQUAL)
Description: CSD-M is a standardized subject diary based on expert consensus and qualitative subject input to retrieve patient reported subjective sleep parameters related to the prior night's sleep. Sleep quality (sQUAL) and how well rested subjects felt at awaking are rated on a 5-point Likert scale ranging from 1 (very poor) to 5 (very good). Higher ratings indicate better sleep quality and more refreshing/restorative quality of sleep (sFRESH). CSD-M parameters analyzed includes: sFRESH and sQUAL. Positive change in sFRESH and sQUAL indicates improvement.
Time Frame: Day 14 to Day 17
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 63 | 58 | 57 | 56 | 58
Units on a Scale
  sFRESH | 0.13 (1.085) [lower limit 1.085] | 0.17 (1.011) [lower limit 1.011] | 0.04 (1.017) [lower limit 1.017] | 0.11 (1.073) [lower limit 1.073] | -0.03 (0.898) [lower limit 0.898]
  sQUAL | 0.19 (1.242) [lower limit 1.242] | 0.24 (1.129) [lower limit 1.129] | -0.07 (1.083) [lower limit 1.083] | 0.02 (1.120) [lower limit 1.120] | -0.12 (1.010) [lower limit 1.010]

45. Secondary Outcome: Change in Subjective Sleep Parameters From Day 14 as Compared to Day 17 Using Consensus Sleep Diary-Morning Administration (CSD-M): Number of Nighttime Awakenings (s-nNAW)
Description: CSD-M is a standardized participant diary based on expert consensus and qualitative participant input to retrieve patient reported subjective sleep parameters related to the prior night's sleep. Higher ratings indicate better sleep quality and more refreshing/restorative quality of sleep. CSD-M parameters analyzed includes: s-nNAW. Negative change in s-nNAW indicate improvement.
Time Frame: Day 14 to Day 17
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 63 | 58 | 57 | 56 | 58
awakenings | 0.16 (3.525) [lower limit 3.525] | -0.59 (2.009) [lower limit 2.009] | -0.35 (1.217) [lower limit 1.217] | -0.36 (1.052) [lower limit 1.052] | -0.34 (1.396) [lower limit 1.396]

46. Secondary Outcome: Number of Participants With Withdrawal Symptoms of JNJ-42847922 as Measured by Physician Withdrawal Checklist (PWC) From Day 14 to Day 17
Description: PWC-20 is a reliable, sensitive instrument having 20-items used to assess potential withdrawal symptoms following cessation of treatment. Items are as follows: Loss of Appetite, Nausea-Vomiting, Diarrhea, Anxiety-Nervousness, Irritability, Dysphoric Mood-Depression, Insomnia, Fatigue, Poor Coordination, Restlessness, Diaphoresis, Tremor, Dizziness, Headaches, Stiffness, Weakness, Increased Acuity Sound Smell Touch (IASST), Paresthesias, Remember, Derealization. Each item score ranges from 0 (not present)-3 (severe), where higher scores = more affected condition. Total score ranges from 0-60, where higher score indicates more affected condition. PWC-20 score was imputed as follows: sum of the non-missing items * (total number of items) / (number of items non-missing).
Time Frame: Day 14 to Day 17
Population: SAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure. 1 participant who was randomized to JNJ-42847922 10 mg dose group received 5 mg of JNJ-42847922 and was summarized under 5 mg dose group for safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 69 | 69 | 70 | 68 | 69
Participants
  Loss of Appetite: No Symptoms | 65 | 69 | 65 | 68 | 66
  Loss of Appetite: Improved Symptoms | 0 | 0 | 4 | 0 | 1
  Loss of Appetite: Symptoms Present and Unchanged | 0 | 0 | 0 | 0 | 0
  Loss of Appetite: New or Worsened Symptoms | 4 | 0 | 1 | 0 | 2
  Nausea-Vomiting: No Symptoms | 67 | 67 | 66 | 67 | 63
  Nausea-Vomiting: Improved Symptoms | 0 | 1 | 3 | 0 | 5
  Nausea-Vomiting: Symptoms Present and Unchanged | 0 | 0 | 0 | 0 | 1
  Nausea-Vomiting: New or Worsened Symptoms | 2 | 1 | 1 | 1 | 0
  Diarrhea: No Symptoms | 65 | 69 | 67 | 67 | 63
  Diarrhea: Improved Symptoms | 2 | 0 | 1 | 1 | 4
  Diarrhea: Symptoms Present and Unchanged | 0 | 0 | 1 | 0 | 0
  Diarrhea: New or Worsened Symptoms | 2 | 0 | 1 | 0 | 2
  Anxiety-Nervousness: No Symptoms | 64 | 68 | 64 | 62 | 62
  Anxiety-Nervousness:Improved Symptoms | 2 | 1 | 3 | 3 | 5
  Anxiety-Nervousness:Symptoms Present and Unchanged | 2 | 0 | 1 | 2 | 0
  Anxiety-Nervousness: New or Worsened Symptoms | 1 | 0 | 2 | 1 | 2
  Irritability: No Symptoms | 58 | 58 | 59 | 60 | 58
  Irritability:Improved Symptoms | 6 | 9 | 5 | 4 | 9
  Irritability:Symptoms Present and Unchanged | 3 | 1 | 3 | 3 | 0
  Irritability:New or Worsened Symptoms | 2 | 1 | 3 | 1 | 2
  Dysphoric Mood: No Symptoms | 66 | 66 | 68 | 65 | 66
  Dysphoric Mood: Improved Symptoms | 0 | 3 | 1 | 1 | 1
  Dysphoric Mood: Symptoms Present and Unchanged | 2 | 0 | 1 | 1 | 0
  Dysphoric Mood: New or Worsened Symptoms | 1 | 0 | 0 | 1 | 2
  Insomnia: No Symptoms | 12 | 14 | 11 | 17 | 16
  Insomnia: Improved Symptoms | 19 | 15 | 13 | 11 | 15
  Insomnia: Symptoms Present and Unchanged | 27 | 28 | 32 | 28 | 21
  Insomnia: New or Worsened Symptoms | 11 | 12 | 14 | 12 | 17
  Fatigue: No Symptoms | 30 | 43 | 41 | 45 | 44
  Fatigue: Improved Symptoms | 21 | 15 | 19 | 8 | 14
  Fatigue: Symptoms Present and Unchanged | 5 | 7 | 8 | 9 | 5
  Fatigue: New or Worsened Symptoms | 13 | 4 | 2 | 6 | 6
  Poor Coordination: No Symptoms | 61 | 65 | 63 | 61 | 61
  Poor Coordination: Improved Symptoms | 6 | 3 | 7 | 5 | 5
  Poor Coordination: Symptoms Present and Unchanged | 1 | 1 | 0 | 1 | 1
  Poor Coordination: New/Worsened Symptoms | 1 | 0 | 0 | 1 | 2
  Restlessness:No Symptoms | 55 | 59 | 59 | 60 | 60
  Restlessness:Improved Symptoms | 9 | 6 | 9 | 5 | 7
  Restlessness:Symptoms Present and Unchanged | 3 | 2 | 1 | 1 | 1
  Restlessness:New or Worsened Symptoms | 2 | 2 | 1 | 2 | 1
  Diaphoresis:No Symptoms | 64 | 68 | 65 | 65 | 64
  Diaphoresis:Improved Symptoms | 3 | 1 | 2 | 2 | 2
  Diaphoresis:Symptoms Present and Unchanged | 0 | 0 | 0 | 0 | 1
  Diaphoresis:New or Worsened Symptoms | 2 | 0 | 3 | 1 | 2
  Tremor: No Symptoms | 66 | 68 | 69 | 68 | 67
  Tremor: Improved Symptoms | 2 | 0 | 0 | 0 | 0
  Tremor: Symptoms Present and Unchanged | 0 | 1 | 0 | 0 | 0
  Tremor: New or Worsened Symptoms | 1 | 0 | 1 | 0 | 2
  Dizziness:No Symptoms | 63 | 69 | 66 | 64 | 60
  Dizziness: Improved Symptoms | 3 | 0 | 2 | 3 | 7
  Dizziness: Symptoms Present and Unchanged | 1 | 0 | 1 | 1 | 1
  Dizziness:New or Worsened Symptoms | 2 | 0 | 1 | 0 | 1
  Headaches:No Symptoms | 56 | 51 | 61 | 60 | 56
  Headaches:Improved Symptoms | 9 | 12 | 4 | 7 | 3
  Headaches:Symptoms Present and Unchanged | 2 | 5 | 3 | 0 | 3
  Headaches:New or Worsened Symptoms | 2 | 1 | 2 | 1 | 7
  Stiffness:No Symptoms | 59 | 62 | 64 | 63 | 59
  Stiffness:Improved Symptoms | 8 | 2 | 2 | 3 | 3
  Stiffness:Symptoms Present and Unchanged | 1 | 2 | 2 | 0 | 1
  Stiffness:New or Worsened Symptoms | 1 | 3 | 2 | 2 | 6
  Weakness:No Symptoms | 61 | 69 | 65 | 65 | 65
  Weakness:Improved Symptoms | 3 | 0 | 3 | 3 | 2
  Weakness:Symptoms Present and Unchanged | 3 | 0 | 1 | 0 | 0
  Weakness:New or Worsened Symptoms | 2 | 0 | 1 | 0 | 2
  IASST: No Symptoms | 64 | 66 | 66 | 63 | 62
  IASST: Improved Symptoms | 1 | 1 | 1 | 3 | 2
  IASST: Symptoms Present and Unchanged | 2 | 1 | 0 | 0 | 1
  IASST: New or Worsened Symptoms | 2 | 1 | 3 | 2 | 4
  Paresthesias:No Symptoms | 62 | 68 | 66 | 68 | 68
  Paresthesias:Improved Symptoms | 4 | 0 | 2 | 0 | 0
  Paresthesias:Symptoms Present and Unchanged | 1 | 1 | 0 | 0 | 0
  Paresthesias:New or Worsened Symptoms | 2 | 0 | 2 | 0 | 1
  Remember:No Symptoms | 50 | 60 | 56 | 56 | 53
  Remember:Improved Symptoms | 9 | 7 | 9 | 8 | 6
  Remember:Symptoms Present and Unchanged | 5 | 1 | 4 | 1 | 5
  Remember:New or Worsened Symptoms | 5 | 1 | 1 | 3 | 5
  Derealization:No Symptoms | 64 | 68 | 68 | 67 | 68
  Derealization:Improved Symptoms | 4 | 1 | 1 | 1 | 1
  Derealization:Symptoms Present and Unchanged | 0 | 0 | 0 | 0 | 0
  Derealization:New or Worsened Symptoms | 1 | 0 | 1 | 0 | 0

47. Secondary Outcome: Benzodiazepine Withdrawal Symptom Questionnaire (BWSQ) Total Score for Self-Assessment of Withdrawal Symptoms on Day 17
Description: The BWSQ is a 20 symptom self-reported questionnaire to investigate withdrawal symptoms. Total score is the sum of item scores. Total scores can range from 0-40 with higher scores indicating greater severity of symptoms. Participants rated the degree to which they were experiencing each symptom as either "0=No," "1=Yes-moderate" or "2=Yes-severe". The questionnaire had been shown to be reliable and to have acceptable construct validity in assessing withdrawal symptoms.
Time Frame: Day 17
Population: SAS included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. Here, N (number of participant analyzed) signifies number of participants evaluable for this outcome measure. One participant who was randomized to JNJ-42847922 10 mg dose group received 5 mg of JNJ-42847922. This participant was summarized under the 5 mg dose group for safety analyses.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
Number analyzed (Participants) | 58 | 54 | 56 | 51 | 55
Units on a Scale | 1.5 (2.58) | 1.2 (1.90) | 2.0 (3.44) | 1.5 (2.93) | 2.0 (3.10)

ADVERSE EVENTS:
Time Frame: Up to Day 17
Description: Safety analysis set included all participants who were randomly assigned to study drug and received at least 1 dose of study drug. One participant who was randomized to JNJ-42847922 10 mg dose group received 5 mg of JNJ-42847922. This participant was summarized under the 5 mg dose group for safety analyses.
Arm/Group | Placebo | JNJ-42847922 5 mg | JNJ-42847922 10 mg | JNJ-42847922 20 mg | Zolpidem
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/72 | 0/73 | 0/71 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/72 | 0/73 | 1/71 | 1/73
Other Adverse Events (participants affected / at risk) | 22/75 | 16/72 | 10/73 | 13/71 | 21/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=75) | JNJ-42847922 5 mg (N=72) | JNJ-42847922 10 mg (N=73) | JNJ-42847922 20 mg (N=71) | Zolpidem (N=73)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=75) | JNJ-42847922 5 mg (N=72) | JNJ-42847922 10 mg (N=73) | JNJ-42847922 20 mg (N=71) | Zolpidem (N=73)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 5 (5)
Fatigue (General disorders) | 8 (8) | 4 (4) | 3 (3) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Disturbance in Attention (Nervous system disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Headache (Nervous system disorders) | 8 (8) | 7 (8) | 4 (6) | 6 (8) | 8 (10)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 4 (5)
Restlessness (Psychiatric disorders) | 4 (4) | 0 (0) | 2 (2) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT03375203/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT03375203/SAP_001.pdf